CLINICAL TRIAL: NCT04627181
Title: The Role Of IV Iron (Ferric Carboxymaltose) And IM Vitamin B12 (Hydroxycobalamin) Supplementation In The Management Of Anaemic Prevalent Indian Hemodialysis Patients: A Parallel Group, Quadruple Blind, Placebo-Controlled, Pragmatic Randomized Control Trial With 2x2 Factorial Design
Brief Title: Do Iron And Vitamin B12 Injections Given Together, Improve Hemoglobin In Patients On Hemodialysis?
Acronym: ALOHA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christian Medical College, Vellore, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12564 (INTERVEN) 29.01.2020
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2020-11

CONDITIONS: Iron Deficiency Anemia; B12 Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Hydroxocobalamin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of four arms: IV ferric carboxymaltose + placebo, IM hydroxycobalamin + placebo, IV ferric carboxymaltose + IM hydroxycobalamin, placebo + placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FCM + placebo (Experimental): 1. Ferric carboxymaltose: Single dose, 500 mg
  2. Placebo: Single dose
  Interventions: Drug: Ferric carboxymaltose; Drug: Placebo
- B12 + placebo (Experimental): 1. Hydroxycobalamine: Single dose, 1000 mcg
  2. Placebo: Single dose
  Interventions: Drug: Hydroxycobalamin; Drug: Placebo
- FCM +B12 (Experimental): 1. Ferric carboxymaltose: Single dose, 500 mg
  2. Hydroxycobalamine: Single dose, 1000 mcg
  Interventions: Drug: Ferric carboxymaltose; Drug: Hydroxycobalamin
- Placebo + placebo (Placebo Comparator): 1. Placebo: Single dose
  2. Placebo: Single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric carboxymaltose — Single dose of ferric carboxymaltose (Encicarb, Emcure Pharmaceuticals Ltd., Pune, India) 500 mg administered intravenously in 100 ml normal saline over 1 hour via the dialysis blood line immediately following HD
  Arms: FCM + placebo; FCM +B12
Drug: Hydroxycobalamin — Single dose of hydroxycobalamine (Trineurosol Hp, Tridoss Laboratories, Mumbai, India) 1000 mcg administered intramuscularly in the deltoid of the non-fistula arm immediately following HD
  Arms: B12 + placebo; FCM +B12
Drug: Placebo — Single dose of 1 ml of distilled water injected intramuscularly in the deltoid of the non-fistula arm immediately following HD
  Arms: FCM + placebo; Placebo + placebo
Drug: Placebo — Single dose of 100 ml normal saline administered intravenously over 1 hour via the dialysis blood line immediately following HD
  Arms: B12 + placebo; Placebo + placebo

SUMMARY:
A parallel group, quadruple blind, placebo-controlled, randomized control trial with 2x2 factorial design to determine the effect of simultaneous IV ferric carboxymaltose and IM hydroxycobalamin supplementation in anemic Indian HD patients

ELIGIBILITY:
Inclusion Criteria:

* All adult prevalent HD patients on HD for at least 3 months with hemoglobin < 11 g/dL

Exclusion Criteria:

* Blood transfusion, blood loss, infection, surgery or change in haemoglobin by > 1 g/dL in the last 1 month
* Hemoglobinopathy
* Cirrhosis
* Hematological malignancy or myeloproliferative disorder
* HIV, HBV or HCV infection
* Any chronic inflammatory disorder
* IV iron or oral/IM B12 received in the last 3 months
* Severe hyperparathyroidism (intact parathyroid hormone > 1,000 pg/mL)
* Pregnancy
* Age < 18 years
* History of asthma or eczema, any history of drug allergy, including allergy to iron preparations
* History of exposure to chemotherapy or cytotoxic drugs - 5-FU, hydroxyurea, hydroxycarbamide, methotrexate, trimethoprim, colchicine, azathioprine
* History of G-CSF use in the last 1 month
* General anaesthesia with nitrous oxide in the last 1 month

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Mean haemoglobin | 30 days
  Mean haemoglobin measured 30 days after the intervention

SECONDARY OUTCOMES:
Sensitivity and specificity of baseline automated red cell indices, peripheral smear red cell indices, and iron indices for diagnosis of iron deficiency | Baseline
  Sensitivity and specificity of baseline peripheral smear hypochromic RBCs >10%, peripheral smear red blood cell anisocytosis > 10%, percentage hypochromic mature red cells (%HYPOm) >6%, reticulocyte hemoglobin content (CHr) < 30 pg, transferrin saturation (TSAT), and serum ferritin, for the diagnosis of iron deficiency anemia. Iron deficiency anemia is defined by an increase in corrected reticulocyte index (reticulocyte % x hematocrit/40) >1% at 7 days and/or increase in hemoglobin by ≥1 g/dL 30 days after administration of IV FCM in the FCM +placebo arm.
Optimum cutoff for baseline automated red cell indices for the diagnosis of iron deficiency anemia using ROC curve analysis | Baseline
  Optimum cutoff of baseline %HYPOm and CHr for the diagnosis of iron deficiency anemia using ROC curve analysis. Iron deficiency anemia is defined by an increase in corrected reticulocyte index (reticulocyte % x hematocrit/40) >1% at 7 days and/or increase in hemoglobin by ≥1 g/dL 30 days after administration of IV FCM in the FCM +placebo arm.
Sensitivity and specificity of baseline peripheral blood smear hypochromia, peripheral blood smear anisocytosis and automated red cell indices for the diagnosis of iron deficiency anemia in participants with TSAT < 30% and TSAT > =30%. | Baseline
  Sensitivity and specificity of > 10% hypochromic red blood cells on peripheral blood smear, >10% red blood cell anisocytosis on peripheral blood smear, %HYPOm > 6%, and CHr < 30 pg measured at baseline, for the diagnosis of iron deficiency anemia in participants with baseline TSAT < 30% and TSAT > 30% respectively. Iron deficiency anemia is defined by an increase in corrected reticulocyte index (reticulocyte % x hematocrit/40) >1% at 7 days and/or increase in hemoglobin by ≥1 g/dL 30 days after administration of IV FCM in the FCM +placebo arm.
Sensitivity and specificity of baseline peripheral smear neutrophil hypersegmentation and cell population data for the diagnosis of B12 deficiency. | Baseline
  Sensitivity and specificity of baseline peripheral smear neutrophil hypersegmentation (>3 percent of neutrophils with ≥5 lobes or ≥1 neutrophil with ≥6 lobes per 100 neutrophils) and cell population data [mean neutrophil volume > 145 fl or mean monocyte volume > 168 fl] for the diagnosis of B12 deficiency. B12 deficiency is defined as an increase in corrected reticulocyte index > 1% (reticulocyte % x hematocrit/40) at 7 days and/or increase in hemoglobin by ≥1 g/dL 30 days after administration of IM hydroxycobalamin in the B12 + placebo group.
Optimum cutoff of cell population data for the diagnosis of B12 deficiency using ROC curve analysis | Baseline
  Optimum cutoff of baseline mean neutrophil volume and mean monocyte volume for the diagnosis of B12 deficiency using ROC curve analysis. B12 deficiency is defined as an increase in corrected reticulocyte index > 1% (reticulocyte % x hematocrit/40) at 7 days and/or increase in hemoglobin by ≥1 g/dL 30 days after administration of IM hydroxycobalamin in the B12 + placebo group.
Adverse effects of IV ferric carboxymaltose and IM hydroxycobalamin therapy | Day 0
  Any adverse events attributable to the use of IV ferric carboxymaltoise and/or IM hydroxycobalamin

OTHER OUTCOMES:
Exploratory: Sensitivity and specificity of red cell anisochromia on peripheral smear for the diagnosis of iron deficiency anemia | Baseline
  Sensitivity and specificity of red cell anisochromia >=25% on the baseline peripheral smear for the diagnosis of iron deficiency anemia. Iron deficiency anemia is defined by an increase in corrected reticulocyte index (reticulocyte % x hematocrit/40) >1% at 7 days and/or increase in hemoglobin by ≥1 g/dL 30 days after administration of IV FCM in the FCM +placebo arm.
Optimal cutoff of baseline serum methylmalonic acid for the diagnosis of B12 deficiency | Baseline
  Optimal cutoff of baseline serum methylmalonic acid for the diagnosis of B12 deficiency. B12 deficiency is defined as an increase in corrected reticulocyte index > 1% (reticulocyte % x hematocrit/40) at 7 days and/or increase in hemoglobin by ≥1 g/dL 30 days after administration of IM hydroxycobalamin in the B12 + placebo group. B12 deficiency is defined as an increase in corrected reticulocyte index > 1% (reticulocyte % x hematocrit/40) at 7 days and/or increase in hemoglobin by ≥1 g/dL 30 days after administration of IM hydroxycobalamin in the B12 + placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Anna T Valson, MD, DM, Study Director — Christian Medical College, Vellore, India; Rizwan Alam, MD, Principal Investigator — Christian Medical College, Vellore, India
Locations (1):
- Christian Medical College, Vellore, Vellore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (including data dictionaries) will be made available immediately after publication of the trial results for an indefinite time period.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately after publication of the results, for an indefinite period
Access Criteria: IPD will be made available to investigators whose proposed use of the data has been approved by an independent review committee in order to achieve aims in the approved proposal. Proposals should be directed to annavalson@cmcvellore.ac.in. To gain access, data requestors will need to sign a data access agreement. Data will be made available at the third party website.